CLINICAL TRIAL: NCT01662141
Title: Investigation of the Reliability to Measure Cardiac Output by a New Ultrasound Dilution Method in Mechanically Ventilated Children After Pediatric Cardiac Surgery
Brief Title: Measure Cardiac Output Using Ultrasound Dilution in Mechanically Ventilated Children
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TSI-S-COstatus-13A-H; IRB (Other: University Hospital in Lund)
Record Dates: First submitted 2012-08-06; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Post Cardiac Surgery
Keywords: Cardiac output; Perivascular Probe

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The measurement of cardiac output (CO) and hemodynamic pressures are vital for proper management of severely hemodynamic compromised patients. A new ultrasound dilution method (COstatus) for cardiac output measurement has been developed.

DETAILED DESCRIPTION:
The thermodilution technique with a pulmonary artery catheter has been the standard in adult patients for cardiac output measurement. However, using pulmonary artery catheter remains a major clinical problem in children due to technical and size constraints.

COstatus measures changes in blood ultrasound velocity in an extracorporeal AV loop caused by body-temperature isotonic saline injected into the central vein and calculates cardiac output derived from a dilution curve.

ELIGIBILITY:
Inclusion Criteria:

* Children <15 kg admitted to pediatric cardiac surgery for corrective surgery and mechanically ventilated were eligible for the study if parents provided informed consent.

Exclusion Criteria:

* Children with known significant tricuspid or mitral valve regurgitations or if it is detected by the preoperative transesophageal echocardiographic examination.
* Children with persistent severe arrhythmias.
* Children with remaining intracardiac shunts after surgery, which may adversely affect the measurement.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric Patients (< 15) in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Measurement of cardiac output by a new ultrasound dilution method in mechanically ventilated children after pediatric cardiac surgery. | Measurements are made during a patient's stay with insitu catheters. The expected average stay is 3-4 days.
  To compare cardiac outputs measured with this new ultrasound dilution method with flowmetry (perivascular probe) using ultrasound transit time measured directly on the aorta in children < 15 kg of weight. Also to assess reliability of COstatus measurements in pediatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lindberg, MD, PhD, Principal Investigator — University Hospital in Lund
Locations (1):
- Children Hospital, BUS, BIVA, Lund, Sweden

REFERENCES:
- [Background] Krivitski NM, Kislukhin VV, Thuramalla NV. Theory and in vitro validation of a new extracorporeal arteriovenous loop approach for hemodynamic assessment in pediatric and neonatal intensive care unit patients. Pediatr Crit Care Med. 2008 Jul;9(4):423-8. doi: 10.1097/01.PCC.0b013e31816c71bc. PMID 18496416